CLINICAL TRIAL: NCT00506688
Title: Randomized, Placebo-controlled, Double-blinded Study to Investigate the Efficacy and Safety of a 24-week Inhalation Treatment With Glutathione in Cystic Fibrosis Patients
Brief Title: Efficacy and Safety Study of Inhaled Glutathione in Cystic Fibrosis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mukoviszidose Institut gGmbH (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Muko-D-GSH-4; EudraCT-number: 2005-003870-88
Record Dates: First submitted 2007-07-24; First posted 2007-07-25 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: reduced glutathione sodium salt — 646 mg GSH-Na powder per vial to prepare a 4ml solution, twice daily for 24 weeks.
  Other Names: TAD 600
Drug: 0.9% normal saline (control) — 4 ml of a 0.9% normal saline solution (9mg/ml NaCl), twice daily for 24 weeks.

SUMMARY:
The majority of cystic fibrosis (CF) patients die from a progressive pulmonary disease.Airway inflammation plays a major role for the pathogenesis of CF lung disease, and ultimately leads to lung destruction. The release of oxidants during the inflammation process leads to a chronic imbalance of oxidants and antioxidants and may be a central component leading to irreversible lung damage in CF patients. The antioxidant glutathione, which is a naturally occurring tripeptide, is depleted in the extracellular epithelial lining fluid of the CF lung. The elevation of reduced level to normal and also the augmentation of glutathione concentrations above the normal level, as observed in smokers and during defence of Pseudomonas infection, may be desirable to avoid lung damage. Data from pilot studies in humans and animals have indicated that the glutathione concentrations in epithelial lining fluid can be elevated by aerosol application.

The main objective of this trial is to evaluate the effect of a 24-week treatment with inhaled glutathione compared with control inhalations (normal saline) on pulmonary function in adult and pediatric CF patients. Secondary objectives are to determine the effects of inhaled glutathione on inflammatory variables, glutathione levels and free elastase in induced sputum and to evaluate the safety and tolerability of the 24-week treatment with inhaled GSH.

There is considerable hope within the CF community that the addition of anti-oxidative therapy to an already comprehensive program for treating the lungs will decrease morbidity and improve the quality of life for patients with CF.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient, 8 years (pediatric 8 - 17 years inclusive; adult 18 years)
* Confirmed diagnosis of CF (positive sweat chloride, 60 mEq/liter by pilocarpine iontophoresis and/or a genotype with two identifiable mutations consistent with CF accompanied by one or more clinical features with the CF phenotype)
* Patient is able to perform acceptable spirometric maneuvers according to ATS standards
* FEV1 > 40% predicted and < 90% predicted
* The patient is clinically stable fulfilling the following:

No evidence of acute upper or lower respiratory tract infection within 4 weeks of screening.

No pulmonary exacerbation requiring an use of i.v./oral/inhaled antibiotics, or oral corticosteroids within 4 weeks of screening.

FEV1 at Visit 2 is within a range of ± 10% of FEV1 from the Visit 1. (If FEV1 at V2 is not within that range, V2 may be re-scheduled once within 7 days)

* Concomitant or chronic medication is planned to be continued unchanged for the entire study duration
* The patient or the patient's legally acceptable representative is able to give informed consent in accordance with ICH and GCP guidelines and local legislation
* Patient is able to comply with the study visit schedule and willing and able to complete the assessments specified in the protocol.

Exclusion Criteria:

* History of allergy/hypersensitivity (including medication allergy) that is deemed relevant to the trial by the investigator. "Relevance" in this context refers to any increased risk of hypersensitivity reaction to trial medication. (Specific concerns currently identified with respect to the use of inhaled glutathione in allergic patients per se are not existing)
* Concomitant inhaled thiol-containing medications (e.g., inhaled N-acetylcysteine).

Such medication had to be finished at least 2 weeks before the screening visit. Oral N-acetylcysteine may be continued.

* New oral or inhaled thiol-containing medications (e.g., inhaled or oral N-acetylcysteine) throughout the study period.
* Patient with a known relevant substance abuse, including alcohol or drug abuse.
* Pregnant or lactating woman or female patient of child bearing potential who is sexually active and not using a medically approved form of contraception such as oral or injectable contraceptives, intrauterine devices, double-barrier method, contraceptive patch, male partner sterilization or condoms.
* Patient with a documented persistent colonization with B. cepacia (defined as more than one positive culture within the past year).
* Start of a new concomitant or chronic medication for CF within 4 weeks of screening.
* Existing cycling medication regimen without completion of at least 3 cycles prior to the screening visit or the drug cycles of other therapies are not in accordance with the 4-week time-schedule for the single visits of this study
* Clinically relevant diseases or medical conditions other than CF or CF-related conditions that, in the opinion of the investigator, would compromise the safety of the patient or the quality of the data. This includes, but is not limited to, significant hematological, hepatic,renal, cardiovascular, and neurological diseases (diabetic patients may participate if their disease is under good control prior to screening).
* Participation in another study with an investigational drug within one month or 6 halflives(whichever is greater) preceding the screening visit.
* The patient is an employee of the investigator or the institution with direct involvement in the trial or other trials under the direction of the investigator or their members.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2007-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Differences between inhaled glutathione and inhaled normal saline with respect to the area under the curve of FEV1 % predicted (forced expiratory volume in 1 second) within the period from baseline to week 24 (V5, EOT) | 24 weeks

SECONDARY OUTCOMES:
Treatment changes with respect to the variables:Spirometry,Peak flow,quality-of-life,Weight/ height,Percentage of neutrophils/other cell types (induced sputum),Induced sputum levels of glutathione/ inflammatory mediators,Pulmonary exacerbation | 0,4, 12, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Griese, Prof., Principal Investigator — Dr. von Haunersches Kinderspital (University of Munich, Germany)
Locations (14):
- Germany (14):
  - Charité Campus Virchow Klinikum,Klinik für Pädiatrie, Berlin
  - Universitätskinderklinink, Bochum
  - Uniklinik Köln Mukoviszidose Zentrum, Cologne
  - Ruhrlandklinink, Essen
  - CF-Ambulanz/ Universitätsklinikum Essen, Essen
  - CF-Ambulanz Frankfurt, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Gemeinschaftspraxis CF Ambulanz, Hamburg
  - Med. Hochschule Hannover, Hanover
  - MHH Kinderklinik CF-Ambulanz, Hanover
  - Universitätsklinik, Leipzig
  - CF-Amulanz/ Dr.von Haunersches Kinderspital, Munich
  - Klinikum Innenstadt, Medizinische Klinik / Pneumologie, München
  - Clemenshospital GmbH,Akademisches Lehrkrankenhaus der Westfälischen Wildhelms-Universität Münster, Münster

REFERENCES:
- [Derived] Griese M, Kappler M, Eismann C, Ballmann M, Junge S, Rietschel E, van Koningsbruggen-Rietschel S, Staab D, Rolinck-Werninghaus C, Mellies U, Kohnlein T, Wagner T, Konig S, Teschler H, Heuer HE, Kopp M, Heyder S, Hammermann J, Kuster P, Honer M, Mansmann U, Beck-Speier I, Hartl D, Fuchs C; Glutathione Study Group; Hector A. Inhalation treatment with glutathione in patients with cystic fibrosis. A randomized clinical trial. Am J Respir Crit Care Med. 2013 Jul 1;188(1):83-9. doi: 10.1164/rccm.201303-0427OC. PMID 23631796